CLINICAL TRIAL: NCT02516319
Title: A Feasibility Study to Determine an Adequate Dose of ICG for the Liver Function Assessment System in Healthy Volunteers
Brief Title: Liver Function Assessment - Feasibility and Dosing Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to discontinue product development.
Sponsor: Cardiox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LFA-0001
Record Dates: First submitted 2015-07-21; First posted 2015-08-05 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Hepatic Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Serial Blood Draws (Active Comparator): Cohorts 3 and 4 - weight based doses of ICG dye followed by serial blood draws at 5, 10, 15 and 20 minutes post ICG injection.
  Interventions: Drug: ICG Dye
- Liver Funtion Test Dye Detection Monitor (Experimental): All cohorts receive continuous LFT monitoring post ICG injection.
  Interventions: Drug: ICG Dye

INTERVENTIONS:
Drug: ICG Dye

SUMMARY:
The purpose of this study is to 1) determine the feasibility of using Cardiox Liver Function Assessment System (LFA) to measure indocyanine green (ICG) clearance; 2) determine an adequate dose based on LFA technology and 3) determine an adequate time period for LFA determination.

DETAILED DESCRIPTION:
Four cohorts of subjects will be enrolled. The fist two cohorts will receive fixed doses of ICG dye (2.5 mg, 5.0 mg, 7.5 mg, 10.0 mg) followed by 20 minutes of LFT monitoring. The final two cohorts will receive weight based doses of ICG dye (0.1 mg/kg, 0.5 mg/kg) followed by 20 minutes of LFT monitoring. Additionally the final two cohorts will have serial blood draws before the ICG dose and at 5, 10, 15 and 20 minutes post ICG dose.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 to 75 years, inclusive
* Informed consent documentation understood and signed.

Exclusion Criteria:

* Known allergy or sensitivity to the ICG or to iodide contrast dye
* Pregnant women or those nursing babies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
ICG dye detection using the LFT system compared to serial blood sampling ethods. | 20 minutes post ICG dose
  Determination of an adequate dose for the Cardiox Liver Functioning Assessment LFA system to produce liver function assessments consistent with serial blood sampling methods.

SECONDARY OUTCOMES:
ICG fluorescence detection at the scaphoid fossa of the ears | 20 minutes post ICG dose
Repeatability of the Cardiox LFA system to detect the ICG fluorescence in the same subjects over time. | 20 minutes post ICG dose

OTHER OUTCOMES:
Adverse-event recording | Two hours post ICG dose
Physical Examination | Up to one hour post ICG dose
Blood pressure | Up to one hour post ICG dose
Heart rate | Up to one hour post ICG dose
Respiration | Up to one hour post ICG dose

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Jopling, M.D, Principal Investigator — Cardiox Corporation